CLINICAL TRIAL: NCT00221663
Title: Clinical Trial Comparing a Conventional Median Sternotomy Versus a Minimally Invasive Technique for Aortic Valvular Replacement in Adults
Brief Title: Conventional Versus Mini-Sternotomy for Aortic Valve Surgery
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Jean Pierre LEROY, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 7945-00; 2000-05
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2008-08-15 (Estimated); Status verified 2008-08

CONDITIONS: Heart Valve Diseases
Keywords: Cardiac surgery; Aortic valve replacement; Minimally invasive surgery; Perioperative course
MeSH Terms: conditions — Heart Valve Diseases | interventions — Sternotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: surgery techniques (sternotomy for aortic valve replacement)

SUMMARY:
Minimally-invasive operative techniques have been introduced in cardiac surgery. These techniques may have several advantages such as a decrease in post operative pain, lower morbidity and mortality, faster recovery, and a shorter hospital stay. However, these advantages have rarely been documented in the setting of a formal randomized controlled trial.

DETAILED DESCRIPTION:
Background:

Minimally invasive techniques for cardiac surgery should be formally evaluated.

Design:

Randomized, single-blind, monocentric trial.

Interventions Compared:

Median sternotomy versus minimally invasive technique.

Eligibility Criteria:

Indication of isolated aortic valvular replacement, preoperative American Society of Anesthesiologists (ASA) class < = 3, left ventricular ejection fraction > = 40%.

Primary Outcome:

Forced expiratory volume and peak expiratory volume/second at 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Indication of isolated aortic valvular replacement
* Preoperative ASA class < = 3
* Left ventricular ejection fraction > = 40%
* Signed informed consent

Exclusion Criteria:

* Aortic or mitral insufficiency > 3
* History of cardiac surgery
* Acute pulmonary edema
* Endocarditis
* Chronic renal insufficiency decompensation
* Operative coagulation disorders regardless of etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2002-01; Primary Completion 2002-01 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume and peak expiratory volume/second | at 48 hours

SECONDARY OUTCOMES:
Forced expiratory volume | at 24 hours
Peak expiratory volume/s at 24 hours
Pro-inflammatory cytokines on tracheal aspiration samples
Transfusion requirements during the first 24 hours post operative
Hemodynamic parameters
Duration of surgery extracorporeal circulation (ECC) and aortic-cross-clamp-time
Consumption of analgetics
Morbidity and mortality during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Janvier, Pr, Principal Investigator — University Hospital, Bordeaux; Joachim Calderon, Dr, Principal Investigator — University Hospital, Bordeaux France; Geneviéve Chene, Pr, Study Chair — University Hospital, Bordeaux France
Locations (1):
- Hôpital Cardiologique du Haut Lévêque, Pessac, France